CLINICAL TRIAL: NCT02818244
Title: Accuracy of Commercially Available Heart Rate Monitors II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Marc Gillinov, MD, Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 16-743
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: commercial heart monitors; accuracy; EKG; varying degrees of exertion
MeSH Terms: interventions — Heart Rate Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Fit Bit Blaze (Active Comparator): Fit Bit Blaze Heart Rate Monitoring Device
  Interventions: Device: Fit Bit Blaze Heart Rate Monitoring Device
- Garmin Forerunner 235 (Active Comparator): Garmin Forerunner 235 Heart Rate Monitoring Device
  Interventions: Device: Garmin Forerunner 235 Heart Rate Monitoring Device
- Tom Tom Spark Cardio (Active Comparator): Tom Tom Spark Cardio Heart Rate Monitoring Device
  Interventions: Device: Tom Tom Spark Cardio Heart Rate Monitoring Device
- Apple Watch (Active Comparator): Apple Watch Heart Rate Monitoring Device
  Interventions: Device: Apple Watch Heart Rate Monitoring Device
- Scosche Rhythm + (Active Comparator): Scosche Rhythm + Heart Rate Monitoring Device
  Interventions: Device: Scosche Rhythm + Heart Rate Monitor

INTERVENTIONS:
Device: Fit Bit Blaze Heart Rate Monitoring Device
  Arms: Fit Bit Blaze
Device: Garmin Forerunner 235 Heart Rate Monitoring Device
  Arms: Garmin Forerunner 235
Device: Tom Tom Spark Cardio Heart Rate Monitoring Device
  Arms: Tom Tom Spark Cardio
Device: Apple Watch Heart Rate Monitoring Device
  Arms: Apple Watch
Device: Scosche Rhythm + Heart Rate Monitor
  Arms: Scosche Rhythm +

SUMMARY:
In 2015, over 85 million fitness wearables were sold worldwide and the market is projected to expand to 110 million units sold in 2017. Of all wearable technology, fitness devices that track heart rate are predicted to be the most popular. At the elite level, commercial heart rate monitors are being used by athletes like LeBron James, Blake Griffin, and Matthew Dellavedova to monitor and alter their behaviors for peak athletic performance. Millions of ordinary consumers purchase fitness trackers that include heart rate monitors in order to help them to maintain their health and wellness. As popularity of these fitness devices grows, assessment of the accuracy of heart rate measurements becomes increasingly important.

DETAILED DESCRIPTION:
In a previous trial, investigators compared the accuracy of four devices (Apple Watch, Fitbit Charge HR, Mio Fuse, Basis Peak) worn by subjects while performing a graded exercise program on a treadmill. Investigators discovered that the Apple Watch and Mio Fuse had a correlation coefficient (rc) of .91, Fitbit Charge HR had an rc of .84, and Basis Peak had an rc of .83. That study has been submitted for publication.

Reviewers of the first study raised an important question: how do commercial optical heart rate monitors perform when measuring heart rate during other popular forms of exercise? This study addresses that question.

Objective:

The objective of this study is to evaluate the accuracy of four heart rate monitors when used during three different exercises: treadmill, stationary bicycle, elliptical trainer.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able and willing to exercise for a total of fifteen minutes

Exclusion Criteria:

* Health issues that preclude or contraindicate walking and/or jogging, including cardiovascular, orthopedic, pulmonary and other conditions
* Presence of a cardiac pacemaker
* Known cardiovascular disease
* Known heart rhythm disorders
* Use of Beta-blockers or antiarrhythmic medications
* Tattoos around the wrist or forearm area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gillinov, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects who met inclusion criteria and had no exclusions were enrolled. All subjects who were consented, participated and completed the study wearing a device on each wrist.
Units Other Than Participants: Heart Rate Monitors
Groups:
- Fit Bit Blaze: Fit Bit Blaze Heart Rate Monitoring Device Standard ECG Polar Chest strap Scosche Rhythm+
- Garmin Forerunner 235: Garmin Forerunner 235 Heart Rate Monitoring Device Standard ECG Polar Chest strap Scosche Rhythm+
- Tom Tom Spark Cardio: Tom Tom Spark Cardio Heart Rate Monitoring Device Standard ECG Polar Chest strap Scosche Rhythm+
- Apple Watch: Apple Watch Heart Rate Monitoring Device Standard ECG Polar Chest strap Scosche Rhythm+
Period: Overall Study
Arm/Group | Fit Bit Blaze | Garmin Forerunner 235 | Tom Tom Spark Cardio | Apple Watch
Started | 25; 25 Heart Rate Monitors | 25; 25 Heart Rate Monitors | 25; 25 Heart Rate Monitors | 25; 25 Heart Rate Monitors
Completed | 25; 25 Heart Rate Monitors | 25; 25 Heart Rate Monitors | 25; 25 Heart Rate Monitors | 25; 25 Heart Rate Monitors
Not Completed | 0; 0 Heart Rate Monitors | 0; 0 Heart Rate Monitors | 0; 0 Heart Rate Monitors | 0; 0 Heart Rate Monitors

BASELINE CHARACTERISTICS:
Units Other Than Participants: Heart Rate
Groups:
- Fit Bit Blaze: Fit Bit Blaze Heart Rate Monitoring Device Monitoring Device Standard ECG Polar Chest strap Scosche Rhythm+
- Garmin Forerunner 235: Garmin Forerunner 235 Heart Rate Monitoring Device Monitoring Device Standard ECG Polar Chest strap Scosche Rhythm+
- Tom Tom Spark Cardio: Tom Tom Spark Cardio Heart Rate Monitoring Device Monitoring Device Standard ECG Polar Chest strap Scosche Rhythm+
- Apple Watch: Apple Watch Heart Rate Monitoring Device Monitoring Device Standard ECG Polar Chest strap Scosche Rhythm+
- Total: Total of all reporting groups
Arm/Group | Fit Bit Blaze | Garmin Forerunner 235 | Tom Tom Spark Cardio | Apple Watch | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Number analyzed (Heart Rate) | 25 | 25 | 25 | 25 | 100
Age, Categorical [Count of Units; unit: Heart Rate]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 25 | 100
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Units; unit: Heart Rate]
  Female | 14 | 12 | 15 | 13 | 54
  Male | 11 | 13 | 10 | 12 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
    (all) |  |  |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure: Heart Rate Monitor Accuracy Compared to ECG Expressed as Correlation Coefficient.
Description: The primary outcome measure is the accuracy of each heart rate monitor compared to ECG. This will be expressed by the correlation coefficient and will also be depicted by Bland-Altman plots.
Time Frame: 24 minutes
Measure: Mean (95% Confidence Interval); unit: Concordance Correlation Coefficient wECG
Arm/Group | Fit Bit Blaze | Garmin Forerunner 235 | Tom Tom Spark Cardio | Apple Watch
Number analyzed (Participants) | 25 | 25 | 25 | 25
Concordance Correlation Coefficient wECG | .67 [.615 to .719] | .81 [.776 to .843] | .83 [.799 to .860] | .92 [.903 to .934]

ADVERSE EVENTS:
Time Frame: 24 minutes
Arm/Group | Fit Bit Blaze | Garmin Forerunner 235 | Tom Tom Spark Cardio | Apple Watch
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes